CLINICAL TRIAL: NCT04860115
Title: Impact of Novel Thoracic Wall Blocks With Dexmetomidine on Inflammatory Markers Following Breast Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Elizabeth Cancer Institute, Slovakia (Other)
Collaborators: F.D. Roosevelt Teaching Hospital with Policlinic Banska Bystrica (Other); Louis Pasteur University Hospital Kosice (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-2021/EK OUSA
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Inflammatory Markers
Keywords: PEC II; PIFB; breast cancer; NLR
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: 120 patients randomized into two groups of 60 patients. Group B (PECS II+PIFB with dexmetomidine) and Group C (control).
Who Masked: Participant, Outcomes Assessor
Masking Description: Intervention will be done under general anesthesia so participant will be blinded and primary outcome which will be laboratory test will be assessed by a person not aware of intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block group (Experimental): Patients in a Block group will be anesthetized and receive PECS II+PIFB with dexmetomidine prior to their surgery.
  Interventions: Procedure: Modified pectoralis block (PEC II) and pecto-intercostal fascial plane block (PIFB)
- Control group (No Intervention): Patients in a Control group will receive a standard general anesthesia the same way as patients in the interventional group but without regional anesthesia.

INTERVENTIONS:
Procedure: Modified pectoralis block (PEC II) and pecto-intercostal fascial plane block (PIFB) — PECS II: Ultrasound guided block involving injection of 20 ml of 0.25% L-bupivacaine with dexmetomidine into an interfascial plane between the serratus anterior muscle and the external intercostal muscles followed by the needle withdrawal into an interfascial plane between the pectoralis major and pectoralis minor muscle where further 10ml will be administered.
  PIFB: Ultrasound guided block involving injection of 10 ml of 0.25% L-bupivacaine with dexmetomidine into an iterfascial plane between the pectoralis major and the intercostal muscles approximately 2 cm laterally from the sternum to cover T2 to T6 dermatomes.
  Arms: Block group

SUMMARY:
The study will test the hypothesis that inflammatory markers measured at 24 hours after breast cancer surgery will be lower in patients receiving PECS II and PIFB blocks, supplemented with dexmetomidine compared to standard care group.

DETAILED DESCRIPTION:
Breast cancer is a devastating disease. Surgery is the mainstay of treatment which can lead to ongoing patient difficulties. Severe acute pain after surgery is one of major risk factors for developing persistent postsurgical pain. Subsequent physiological stress caused by this severe pain may negatively influence the immune response leading to a worse prognosis.

Regional anesthesia is very effective in management of peri- and postoperative pain. Epidural block, paravertebral block and intercostal nerve blocks have been proven over time to be effective in preventing postoperative pain. However, their widespread use has been hampered by technical difficulty and inherent risks.

Unlike the aforementioned blocks, novel thoracic wall blocks, namely modified pectoralis block (PECS II) and pecto-intercostal fascial block (PIFB) are safe, simple and effective.

Efforts to prolong and improve analgesia following single shot blocks has led to the introduction of adjuvants into the local anesthetic. Dexmetomidine is a superselective Alpha 2 agonist with a proven ability to prolong the duration of neuraxial, peripheral nerve and interfascial plane blocks.

Chronic inflammation is recognized as a risk factor for initiation, progression and further spread of malignant growth. Surgical insult leads to inflammatory response which facilitates the development of a metastatic disease. Many inflammatory markers were proven to be independent prognostic factors in breast cancer patients.

The investigators propose to study the impact of novel thoracic wall blocks with dexmetomidine on simple inflammatory markers obtained from full blood count (NLR, PLR, NPR, PDW, MPV, RDW) after breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with ductal carcinoma (stage 1 to 3) undergoing primary potentially curative unilateral mastectomy.
* Older than 18 years
* ASA I-III

Exclusion Criteria:

* Weight < 50 kg
* BMI > 35
* Allergy to local anaesthetic or dexmetomidine
* Contraindications to NSAIDs use
* Local infection over block site
* Coagulopathy
* Preexisting chronic pain
* Pregnancy
* Autoimmune disease
* Inability to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Difference in NLR | 24 hours after surgery
  Difference in neutrophil-lymphocyte ratio (NLR) between the intervention group and the standard care group measured at 24 hours after breast cancer surgery

SECONDARY OUTCOMES:
Markers of inflammation | 24 hours after surgery
  Difference in Δ NLR, PLR, NPR, PDW, MPV and RDW between the intervention group and the standard care group measured at 24 hours after breast cancer surgery
Intraoperative opioids | Duration of surgery
  Intraoperative consumption of opioids
Pain after surgery | 1,6,12,18,24 hours after surgery
  Numeric rating scale for pain (NRS, 0-10, where 0 means no pain and 10 the worst pain) at 0, 1h, 6h, 12h,18h,24h after surgery at rest and at ipsilateral arm abduction
Opioid consumption | 24 hours
  Total opioid consumption after surgery at 24 h

OTHER OUTCOMES:
Adverse effects | 24 hours
  Incidence of potential adverse effects
Postsurgical pain | 3 months after surgery
  Incidence of postsurgical pain at 1month, 2month and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Hitka, MD, Principal Investigator — St. Elizabeth Cancer Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2016. CA Cancer J Clin. 2016 Jan-Feb;66(1):7-30. doi: 10.3322/caac.21332. Epub 2016 Jan 7. PMID 26742998
- [Background] Fecho K, Miller NR, Merritt SA, Klauber-Demore N, Hultman CS, Blau WS. Acute and persistent postoperative pain after breast surgery. Pain Med. 2009 May-Jun;10(4):708-15. doi: 10.1111/j.1526-4637.2009.00611.x. Epub 2009 Apr 22. PMID 19453965
- [Background] Andersen KG, Kehlet H. Persistent pain after breast cancer treatment: a critical review of risk factors and strategies for prevention. J Pain. 2011 Jul;12(7):725-46. doi: 10.1016/j.jpain.2010.12.005. Epub 2011 Mar 24. PMID 21435953
- [Background] Lee SK, Choi MY, Bae SY, Lee JH, Lee HC, Kil WH, Lee JE, Kim SW, Nam SJ. Immediate postoperative inflammation is an important prognostic factor in breast cancer. Oncology. 2015;88(6):337-44. doi: 10.1159/000368985. Epub 2015 Feb 25. PMID 25721153
- [Background] Duff S, Connolly C, Buggy DJ. Adrenergic, Inflammatory, and Immune Function in the Setting of Oncological Surgery: Their Effects on Cancer Progression and the Role of the Anesthetic Technique in their Modulation. Int Anesthesiol Clin. 2016 Fall;54(4):48-57. doi: 10.1097/AIA.0000000000000120. No abstract available. PMID 27648890
- [Background] Freise H, Van Aken HK. Risks and benefits of thoracic epidural anaesthesia. Br J Anaesth. 2011 Dec;107(6):859-68. doi: 10.1093/bja/aer339. Epub 2011 Nov 4. PMID 22058144
- [Background] Klein SM, Bergh A, Steele SM, Georgiade GS, Greengrass RA. Thoracic paravertebral block for breast surgery. Anesth Analg. 2000 Jun;90(6):1402-5. doi: 10.1097/00000539-200006000-00026. PMID 10825328
- [Background] Kolawole IK, Adesina MD, Olaoye IO. Intercostal nerves block for mastectomy in two patients with advanced breast malignancy. J Natl Med Assoc. 2006 Mar;98(3):450-3. PMID 16573313
- [Background] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Background] de la Torre PA, Garcia PD, Alvarez SL, Miguel FJ, Perez MF. A novel ultrasound-guided block: a promising alternative for breast analgesia. Aesthet Surg J. 2014 Jan 1;34(1):198-200. doi: 10.1177/1090820X13515902. No abstract available. PMID 24396082
- [Background] Kulhari S, Bharti N, Bala I, Arora S, Singh G. Efficacy of pectoral nerve block versus thoracic paravertebral block for postoperative analgesia after radical mastectomy: a randomized controlled trial. Br J Anaesth. 2016 Sep;117(3):382-6. doi: 10.1093/bja/aew223. PMID 27543533
- [Background] Marhofer P, Brummett CM. Safety and efficiency of dexmedetomidine as adjuvant to local anesthetics. Curr Opin Anaesthesiol. 2016 Oct;29(5):632-7. doi: 10.1097/ACO.0000000000000364. PMID 27258154
- [Background] Fritsch G, Danninger T, Allerberger K, Tsodikov A, Felder TK, Kapeller M, Gerner P, Brummett CM. Dexmedetomidine added to ropivacaine extends the duration of interscalene brachial plexus blocks for elective shoulder surgery when compared with ropivacaine alone: a single-center, prospective, triple-blind, randomized controlled trial. Reg Anesth Pain Med. 2014 Jan-Feb;39(1):37-47. doi: 10.1097/AAP.0000000000000033. PMID 24317234
- [Background] Xu L, Hu Z, Shen J, McQuillan PM. Efficacy of US-guided transversus abdominis plane block and rectus sheath block with ropivacaine and dexmedetomidine in elderly high-risk patients. Minerva Anestesiol. 2018 Jan;84(1):18-24. doi: 10.23736/S0375-9393.17.11538-5. Epub 2017 May 19. PMID 28528536
- [Background] Hanahan D, Weinberg RA. Hallmarks of cancer: the next generation. Cell. 2011 Mar 4;144(5):646-74. doi: 10.1016/j.cell.2011.02.013. PMID 21376230
- [Background] Koh CH, Bhoo-Pathy N, Ng KL, Jabir RS, Tan GH, See MH, Jamaris S, Taib NA. Utility of pre-treatment neutrophil-lymphocyte ratio and platelet-lymphocyte ratio as prognostic factors in breast cancer. Br J Cancer. 2015 Jun 30;113(1):150-8. doi: 10.1038/bjc.2015.183. Epub 2015 May 28. PMID 26022929
- [Background] Krenn-Pilko S, Langsenlehner U, Thurner EM, Stojakovic T, Pichler M, Gerger A, Kapp KS, Langsenlehner T. The elevated preoperative platelet-to-lymphocyte ratio predicts poor prognosis in breast cancer patients. Br J Cancer. 2014 May 13;110(10):2524-30. doi: 10.1038/bjc.2014.163. Epub 2014 Mar 27. PMID 24675383
- [Background] Hu L, Li M, Ding Y, Pu L, Liu J, Xie J, Cabanero M, Li J, Xiang R, Xiong S. Prognostic value of RDW in cancers: a systematic review and meta-analysis. Oncotarget. 2017 Feb 28;8(9):16027-16035. doi: 10.18632/oncotarget.13784. PMID 27926498
- [Result] Ni Eochagain A, Burns D, Riedel B, Sessler DI, Buggy DJ. The effect of anaesthetic technique during primary breast cancer surgery on neutrophil-lymphocyte ratio, platelet-lymphocyte ratio and return to intended oncological therapy. Anaesthesia. 2018 May;73(5):603-611. doi: 10.1111/anae.14207. Epub 2018 Feb 19. PMID 29457215